CLINICAL TRIAL: NCT03585920
Title: The Influence of Fat Perception on Satiety From Consumption of Reduced Fat Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: University of Sussex (Other); Quadram Institute Bioscience (Other); Unilever R&D (Industry); PepsiCo Global R&D (Industry); Mondelēz International, Inc. (Industry); Arla Foods (Industry); Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Lisa Methven, Associate Professor in Food and Sensory Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UREC 18/05
Record Dates: First submitted 2018-06-14; First posted 2018-07-13 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Appetitive Behavior; Individual Difference; Food Sensitivity; Food Preferences
Keywords: Fat; Oral sensitivity; Appetite; Metabolism
MeSH Terms: conditions — Appetitive Behavior; Food Intolerance; Food Preferences; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: This is a 3 way crossover design using a pre-load study protocol that is standard for behavioural appetite studies. The study will be conducted single-blind, as it is not feasible to blind the researcher to the pre-load food products. Each participant will attend 3 visits, the pre-load study foods will be presented to them with random blinding codes.
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Control (standard fat) (Active Comparator): Expanded Corn Snack. Positive control (13 g oil per 40 g snack portion)
  Interventions: Behavioral: Expanded Corn Snack
- Negative Control (reduced fat) (Experimental): Expanded Corn Snack. Negative control (<8 g oil per 40 g snack)
  Interventions: Behavioral: Expanded Corn Snack
- Reduced Fat Sensory Matched (Experimental): Expanded Corn Snack. Reduced fat optimised (<8 g oil, matched sensory signals)
  Interventions: Behavioral: Expanded Corn Snack

INTERVENTIONS:
Behavioral: Expanded Corn Snack — A standard expanded snack will be used in each of the 3 arms, the content and type of fat added to the snack is varied in the two experimental arms.

SUMMARY:
The present study aims to investigate the effect of fat level and fat type of a snack on self-reported satiety and associated biomarkers. The relevant individual differences will also be investigated.

DETAILED DESCRIPTION:
The aims are: (1) To determine whether reducing fat in a snack leads to rebound hunger and higher food intake at the subsequent meal, (2)To determine whether a low fat snack product matched for expected satiety leads to differences in post-ingestive satiety (i.e. mouth-gut discordance), (2) To determine whether individual differences in sensory perception influence expected or post-ingestive satiety.

Stage 1, Characterising Volunteers:

Fat is perceived through three sensory modalities; mouthfeel, taste and odour. Humans vary in their perception of fat across all sensory modalities. Volunteers will be characterised on their ability to taste fatty acids and perceive mouthfeel.

Stage 2, Establish Sensory Tolerance in Expected Satiety of a fat reduced snack model:

Reduced fat products are typically reformulated to match the perceived texture and mouthfeel of the original product. This stage aims to quantify sensory tolerance to fat reduction.

Stage 3, Establish Mouth Gut Discordance of a fat reduced snack model:

Using a standard preload study design, and the same fat-emulsion snack model from stage 2, the investigators will contrast effects of 3 test samples in a balanced cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18-70 years
* Body mass index (BMI): 18-32 kg/m2
* Fasting glucose < 7 mmol/l
* Fasting total cholesterol < 7.5 mmol/L
* Fasting triglycerides < 2.3 mmol/L
* Weight stable in the last three months

Exclusion Criteria:

* Diagnosed with diabetes or cardiovascular disease (e.g. stroke or heart attack), gastrointestinal (e.g. Irritable bowel syndrome (IBS), inflammatory conditions, gastroenteritis), endocrine or renal diseases
* Smoker
* Taking prescribed medications that could influence study outcomes (e.g. lipid lowering medications, anti-depressants, anticoagulants)
* Food allergies (e.g. gluten, dairy) and intolerances (e.g. lactose)
* Drug abuse
* Anaemia (men: haemoglobin<130 g/L and women <115 g/L)
* Hypertension (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
* Planning or currently on a weight reducing programme
* Pregnancy, planned pregnancy in the next year or lactating
* Currently taking part or participation in other research studies within the last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Food Intake (gram) | One measurement taken at 240 min after start of each stage 3 visit day.
  Weighed food intake (gram) at ad libitum meal

SECONDARY OUTCOMES:
Satiety hormone Cholecystokinin (CCK) | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Cholecystokinin (CCK) is one of the satiety hormones, a peptide hormone of the gastrointestinal system responsible for stimulating the digestion of fat and modulating appetite. Blood sample will be collected in order to analyze the level (pg/ml) of cholecystokinin (CCK).
Satiety hormone Peptide YY (PYY) | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Peptide YY (PYY) is one of the satiety hormones, acting to reduce appetite. Blood sample will be collected in order to analyze the level (pg/ml) of Peptide YY (PYY).
Satiety hormone Glucagon-like peptide-1 (GLP-1) | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Glucagon-like peptide-1 (GLP-1) is one of the satiety hormones, modulating appetite. Blood sample will be collected in order to analyze the level (pg/ml) of Glucagon-like peptide-1 (GLP-1).
Satiety hormone Ghrelin | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Ghrelin is termed as the 'hunger hormone' as it stimulates appetite, increases food intake and promotes fat storage. Blood sample will be collected in order to analyze the level (pg/ml) of Ghrelin.
Satiety hormone Leptin | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Leptin is a hormone that can regulate energy intake and modulate hunger. Blood sample will be collected in order to analyze the level (pg/ml) of Leptin.
Satiety hormone Gastric inhibitory polypeptide (GIP) | Sampled via cannula at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  Gastric inhibitory polypeptide (GIP) can modulate appetite. Blood sample will be collected in order to analyze the level (pg/ml) of Gastric inhibitory polypeptide (GIP).
Saliva Samples | Samples at 0, 15, 105, 125, 155, 180 and 240 min on each stage 3 visit day.
  The level (ppm) of metabolomics (e.g. butyrate, propionate, lactate, acetate and 3-hydroxyisovalerate) in un-stimulated saliva will be analyzed using Nuclear Magnetic Resonance (NMR). As all these metabolomics in saliva can be analysed in one run, this is treated as one outcome.
Urine Samples | One sample at start of study day (0 min) and one sample at start of lunch (180 min) on each stage 3 visit day
  Sample for urinary Nuclear Magnetic Resonance (NMR) metabolic profiles. Spectra will be compared and differences in integrated peak areas compared as AU (arbitrary units)
Satiety Ratings | Over 4 hours at time 0, 120, 150, 180 and 240 min on each stage 3 visit day.
  Satiety Ratings on visual analogue unstructured line scale (from 0 (not at all) to 100 (extremely)). The score obtained from participants only represents the hunger or satiety at that time point, which does not represent "good" or "bad" outcome.
Hunger Ratings | Over 4 hours at time 0, 120, 150, 180 and 240 min on each stage 3 visit day.
  Hunger Ratings on visual analogue unstructured line scale (from 0 (not at all) to 100 (extremely)). The score obtained from participants only represents the hunger or satiety at that time point, which does not represent "good" or "bad" outcome.
Individual differences in sensory perception (fatty acid sensitivity) | Sensory perception measures taken once in stage 1 (in the first visit of the study)
  Volunteers will have been characterised on their ability to taste the emulsions samples with the added fatty acid at the level of 0.016% and 0.11% (weight by weight) in Stage 1 (in the first visit). A discrimination forced choice test will be used, where the participant is asked to state the odd sample out of a set. If they can detect fatty acid in the samples correctly three times, they will be classified as hyper-sensitivity, otherwise they will be classified as hypo-sensitivity.
Individual differences in sensory perception (Mouthfeel Sensitivity) | Sensory perception measures taken once in stage 1 (in the first visit).
  A mouthfeel discrimination test will be carried out using savoury biscuits which are constant in overall fat content but vary in mouthfeel characteristics. Four samples will be prepared varying in mouthfeel and participants will be asked to taste the samples and then rate them for the mouthfeel attributes of Crunchiness, Hardness, Greasiness, on visual analogue structured line scale (from 0 (not at all) to 100 (extremely)).
Individual differences in sensory perception (Tactile sensitivity ) | Sensory perception measures taken once in stage 1 (in the first visit).
  Von Frey filaments will be used to evaluate tactile sensitivity on the tongue, and to relate this to taste sensitivity. Participants will be asked to wear a blindfold, the middle of their tongue is then either stimulated or not stimulated with two Von Frey filaments of 0.008g and 0.02g sizes. The participant responds to say whether they have felt the stimulation and how sure they are (signal sure, signal not sure, no signal sure, no signal not sure). This is repeated 10 times in rapid succession. Responses are analysed using an R-index (%) value which is standard for a signal-noise detection test.
Individual differences in sensory perception (Mouth behaviour test ) | Sensory perception measures taken once in stage 1 (in the first visit).
  A simple short questionnaire will be used, which has been validated in the USA, to categorise people as "Crunchers", "Chewers", "Suckers" and "Smooshers". Whereas "Chewers" tend to chew foods to a fine particle size before swallowing, "Crunchers" rapidly crunch and swallow. This questionnaire has been validated in the United States.
Individual differences in sensory perception (Fungiform papillae (FP) density) | Sensory perception measures taken once in stage 1 (in the first visit).
  In order to determine fungiform papillae density on the tongue, a digital camera will be used to record an image of the number of fungiform papillae in two one cm2 areas of the tongue. A small area of the participant's tongue will be temporarily dyed blue using food colour applied by a cotton wool bud. The tongue will then be blotted dry to remove excess moisture prior to recording a digital image. The blue colour will fade after approximately 1 hour and the extent of the colouration is similar to eating certain coloured sweets (e.g. blue Smarties).The number of the fungiform papillae (FP) density will be counted afterwards and quantified as papillae / cm square.
Individual differences in expected satiety | Expected satiety measures taken once in stage 2 (in the second visit).
  7 snack samples will be presented to subjects in a monadic sequential manner (i.e. one at a time) in a balanced order. After tasting each sample, participants will rate expected satiety ( "If you were to consume a full portion of this product, how full do you think you would feel?"and "How long do you think it would be before you felt hungry again?"). Visual analogue unstructured line scales (from 0 (not at all) to 100 (extremely)) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Science, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unlinked / non-identifiable) data will be useful in a meta-analysis and, hence, sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Zhou X, Shen Y, Parker JK, Kennedy OB, Methven L. Relative Effects of Sensory Modalities and Importance of Fatty Acid Sensitivity on Fat Perception in a Real Food Model. Chemosens Percept. 2016;9:105-119. doi: 10.1007/s12078-016-9211-5. Epub 2016 Jul 11. PMID 27594969
- [Background] Stewart JE, Newman LP, Keast RS. Oral sensitivity to oleic acid is associated with fat intake and body mass index. Clin Nutr. 2011 Dec;30(6):838-44. doi: 10.1016/j.clnu.2011.06.007. Epub 2011 Jul 14. PMID 21757270
- [Background] Lett AM, Norton JE, Yeomans MR. Emulsion oil droplet size significantly affects satiety: A pre-ingestive approach. Appetite. 2016 Jan 1;96:18-24. doi: 10.1016/j.appet.2015.08.043. Epub 2015 Sep 4. PMID 26344811
- [Background] Woodend DM, Anderson GH. Effect of sucrose and safflower oil preloads on short term appetite and food intake of young men. Appetite. 2001 Dec;37(3):185-95. doi: 10.1006/appe.2001.0425. PMID 11895319
- [Background] Yeomans MR, Chambers L. Satiety-relevant sensory qualities enhance the satiating effects of mixed carbohydrate-protein preloads. Am J Clin Nutr. 2011 Dec;94(6):1410-7. doi: 10.3945/ajcn.111.011650. Epub 2011 Oct 26. PMID 22030223
- [Background] Keller KL, Liang LC, Sakimura J, May D, van Belle C, Breen C, Driggin E, Tepper BJ, Lanzano PC, Deng L, Chung WK. Common variants in the CD36 gene are associated with oral fat perception, fat preferences, and obesity in African Americans. Obesity (Silver Spring). 2012 May;20(5):1066-73. doi: 10.1038/oby.2011.374. Epub 2012 Jan 12. PMID 22240721
- [Background] Kulkarni BV, Mattes RD. Lingual lipase activity in the orosensory detection of fat by humans. Am J Physiol Regul Integr Comp Physiol. 2014 Jun 15;306(12):R879-85. doi: 10.1152/ajpregu.00352.2013. Epub 2014 Apr 2. PMID 24694384
- [Background] Mennella I, Savarese M, Ferracane R, Sacchi R, Vitaglione P. Oleic acid content of a meal promotes oleoylethanolamide response and reduces subsequent energy intake in humans. Food Funct. 2015 Jan;6(1):204-10. doi: 10.1039/c4fo00697f. Epub 2014 Oct 27. PMID 25347552
- [Background] Jeltema M, Beckley J, Vahalik J. Model for understanding consumer textural food choice. Food Sci Nutr. 2015 May;3(3):202-12. doi: 10.1002/fsn3.205. Epub 2015 Feb 2. PMID 25987995
- [Background] Yackinous C, Guinard JX. Relation between PROP taster status and fat perception, touch, and olfaction. Physiol Behav. 2001 Feb;72(3):427-37. doi: 10.1016/s0031-9384(00)00430-3. PMID 11274688
- [Background] Eldeghaidy S, Marciani L, Hort J, Hollowood T, Singh G, Bush D, Foster T, Taylor AJ, Busch J, Spiller RC, Gowland PA, Francis ST. Prior Consumption of a Fat Meal in Healthy Adults Modulates the Brain's Response to Fat. J Nutr. 2016 Nov;146(11):2187-2198. doi: 10.3945/jn.116.234104. Epub 2016 Sep 21. PMID 27655761

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03585920/Prot_ICF_000.pdf